CLINICAL TRIAL: NCT04099303
Title: A Randomized,Blind, Positive-controlled Phase I Clinical Trial to Preliminary Evaluate the Safety of DTcP Vaccine in Healthy Children Aged Between 2 Months and 6 Years
Brief Title: Phase I Clinical Trial of Diphtheria, Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed .
Acronym: PCTDTcP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CS-CTP-DTcP-Ⅰ
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: Infection; DTcP; Whooping Cough; Vaccine; Diphtheria; Tetanus; Pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Infections | interventions — Tetanus Toxoid; Vaccines, Combined; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Vaccine 1A (Experimental): Subjects received one dose of DTaP aged 4 to 6 years.
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- Vaccine 1B (Active Comparator): Subjects received one dose of DT aged 4 to 6 years.
  Interventions: Biological: Diphtheria and Tetanus Combined Vaccine, Adsorbed
- Vaccine 2A (Experimental): Subjects received one dose of DTcP aged 18 to 24 months.
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- Vaccine 2B (Active Comparator): Subjects received one dose of DTaP aged 18 to 24 months.
  Interventions: Biological: Diphtheria-tetanus-acellular pertussis vaccine
- Vaccine 3A (Experimental): Subjects received three doses of DTcP at 3,4,5 months of age.
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- Vaccine 3B (Active Comparator): Subjects received three doses of DTaP at 3,4,5 months of age.
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed; Biological: Diphtheria-tetanus-acellular pertussis vaccine
- Vaccine 3C (Active Comparator): Subjects received three doses of DTaP-IPV-Hib at 3,4,5 months of age.
  Interventions: Biological: Diphtheria,tetanus,pertussis(acellular,component),poliomyelitis(inactivated) vaccine(absorbed) and Haemophilus influenzae type b conjugate vaccine
- Vaccine 4A (Experimental): Subjects received three doses of DTcP at 2,3,4 months of age.
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed
- Vaccine 4B (Active Comparator): Subjects received three doses of DTaP-IPV-Hib at 2,3,4 months of age.
  Interventions: Biological: Diphtheria,tetanus,pertussis(acellular,component),poliomyelitis(inactivated) vaccine(absorbed) and Haemophilus influenzae type b conjugate vaccine
- Vaccine 4C (Experimental): Subjects received three doses of DTcP at 2,4,6 months of age.
  Interventions: Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed

INTERVENTIONS:
Biological: Diphtheria,Tetanus and Acellular Pertussis (Three Components) Combined Vaccine, Adsorbed — 0.5 mL, Intramuscular Other Name: DTcP
  Arms: Vaccine 1A; Vaccine 2A; Vaccine 3A; Vaccine 3B; Vaccine 4A; Vaccine 4C
Biological: Diphtheria and Tetanus Combined Vaccine, Adsorbed — 2mL, Intramuscular Other Name: DT
  Arms: Vaccine 1B
Biological: Diphtheria-tetanus-acellular pertussis vaccine — 0.5 mL, Intramuscular Other Name: DTaP
  Arms: Vaccine 2B; Vaccine 3B
Biological: Diphtheria,tetanus,pertussis(acellular,component),poliomyelitis(inactivated) vaccine(absorbed) and Haemophilus influenzae type b conjugate vaccine — 0.5 mL, Intramuscular Other Name: PENTAXIM
  Arms: Vaccine 3C; Vaccine 4B

SUMMARY:
Pertussis, diphtheria and tetanus are seriously infectious diseases in children. Since using of the vaccine targeted the three components, it greatly reduced incidence of the three kinds of diseases. The Purpose of this study is to preliminary evaluate the safety of DTcP compared to adsorbed diphtheria and tetanus combined vaccine （DT），Diphtheria-tetanus-acellular pertussis vaccine（DTaP） or PENTAXIM（DTaP-IPV-Hib） in participants.

DETAILED DESCRIPTION:
Study participants will receive a single booster dose of DTcP or a single booster dose of local DT in 4 to 6 years old ,a singel booster dose of DTcP or a single booster dose of DTaP in 18 to 24 months, three basic doses of DTcP or three doses of DTaP/ DTaP-IPV-Hib in 2 to 6 months.Safety profile will be assessed in all subjects up to Day 30 post vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 2months、3months、18-24months and 4-6 years old;
* Willing to provide proof of identity;
* Able to understand and sign the informed consent by guardians or trustees;
* Able and willing comply with the requirements of the protocol by guardians or trustees;
* Subjects of 2 months age have not been vaccinated with diphtheria, IPV, Hib, or 13-valent pneumococcal polysaccharide conjugate vaccine;
* Subjects of 3 months have not been inoculated with vaccines containing diphtheria, Hib, 13-valent pneumococcal polysaccharide conjugate vaccine and Meningococcal Group AC Bivalent Meningococcal Conjugate Vaccine;volunteers of 3 months (C3 group) have not been inoculated with vaccines containing IPV;
* Subjects aged 18-24 months who had completed the immunization program of 3 doses of DTaP and had without the fourth DTaP vaccine ;
* Subjects aged 4-6 years who have completed the immunization program of 4 doses of DTaP or similar vaccines containing DTP component, but who have not received DT vaccine;

Exclusion Criteria:

* Premature birth in infant under 1 year of age (delivery before the 37th week of pregnancy)or low birth weight (birth weight< 2300g for girls,<2500g for boys);
* History of abnormal labor process or asphyxia rescue ;
* Subjects who has a medical history of diphtheria, pertussis or tetanus;
* In the past 30 days, individuals who have had contact with individuals with confirmed pertussis, diphtheria and tetanus diseases in their families;
* Allergic person;
* Any prior administration of blood products in last 3 month;
* Any prior administration of other research medicines in last 1 month;
* Plans to participate in or is participating in any other drug clinical study;
* Any prior administration of attenuated live vaccine in last 14 days;
* Any prior administration of subunit or inactivated vaccines in last 7 days;
* Had fever before vaccination, Subjects with temperature >37.0°C on axillary setting;
* According to the investigator's judgment, the subjects have any other factors that make them unfit to participate in the clinical trial

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-11-25 (Actual)

PRIMARY OUTCOMES:
Safety items of adverse reactions | within 30 minutes post-vaccination
  Occurrence of adverse reactions
Safety items of adverse reactions | within 7 days post-vaccination
  Occurrence of adverse reactions
Safety items of SAE: Occurrence of SAE | within 360 days post-vaccination
  Occurrence of SAE
Safety itmes of laboratory measures: Occurrence of abnormal changes of laboratory measures | the fourth day post-vaccination
  Occurrence of abnormal changes of laboratory measures
Safety items of adverse reactions | within 8-30 days post-vaccination
  Occurrence of adverse reactions
Safety items of adverse reactions | within 30 days post-vaccination
  Occurrence of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yanxia, Principal Investigator — Henan Province Center for Disease Control and Prevention
Locations (1):
- Changge Center for Disease Control and Prevention, Xuchang, Henan, China

IPD SHARING:
Plan to Share IPD: No
In order to maintain the rights of the subject, do not open the IPD